CLINICAL TRIAL: NCT00179725
Title: Phase I/II Open-Label, Dose Escalation Study To Determine The Maximum Tolerated Dose And To Evaluate The Safety Profile of Lenalidomide (Revlimid®) With Liposomal Doxorubicin In Subjects With Advanced Ovarian and Primary Peritoneal Carcinoma
Brief Title: Phase I/II Open-Label, Dose Escalation Study To Determine The Maximum Tolerated Dose And To Evaluate The Safety Profile of Lenalidomide (Revlimid® CC-5013) With Liposomal Doxorubicin In Subjects With Advanced Ovarian and Primary Peritoneal Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-OVRY-001
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2006-04-12 (Estimated); Status verified 2006-04

CONDITIONS: Ovarian Cancer
Keywords: cc-5013; revlimid; ovarian cancer; celgene
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Lenalidomide; liposomal doxorubicin

INTERVENTIONS:
Drug: CC-5013
Drug: liposomal doxorubicin

SUMMARY:
Phase I will determine the MTD and evaluated the safety profile of oral lenalidomide on days 1-21 when given with liposomal doxorubicin on day 1 of every 28 day cycle Phase II will commence once the MTD is established, additional subjects will be enrolled and receive oral lenalidomide on days 1-21 with liposomal doxorubicinon day 1 in 28 day cycles until disease progression is documented.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand and voluntarily sign an informed consent document.
2. Age > or = to 18 years at the time of signing informed consent form.
3. Subjects must be able to adhere to the study visit schedule and other protocol requirements.
4. Histological or cytological documentation of advanced ovarian or primary peritoneal carcinoma.
5. Radiographic or clinical evidence of measurable metastatic advanced ovarian or primary peritoneal carcinoma. Subjects must have measurable disease at least 2 cm in diameter.
6. Subjects must have been treated and progressed following chemotherapy which includes platinum and paclitaxel.
7. ECOG performance status of 0 or 1 (Appendix I: ECOG Performance Status Scale).
8. Must have 2-d Echocardiogram/MUGA indicating a LVEF above the institutional lower limit of normal within 42 days prior to first dose of study drug.

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,500 cells/mm3 (1.5 x 109/L)
   2. Platelet count <100,000 cells/mm3 (100 x 109/L)
   3. Serum creatinine >2.5 mg/dL (221 mmol/L)
   4. Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >1.2 mg/dL (20 mmol/L)
2. Any serious medical condition or psychiatric illness that places the subject at an unacceptable risk for study participation or would prevent the subject from signing the informed consent.
3. Prior history of malignancy (except basal cell or squamous cell carcinoma or carcinoma in situ of the breast) unless the subject has been free of disease for > or = to 1 years.
4. Known brain or leptomeningeal disease (CT scan or MRI of the brain required only in case of clinical suspicion of central nervous system involvement).
5. More than 1 prior chemotherapy regimen. However, subjects with platinum sensitive disease (i.e., subjects who fail a platinum containing regimen at least six months after completing the regimen) who are retreated with a platinum containing regimen are eligible.
6. Concurrent use of any other anti-cancer agents.
7. Any prior use of Lenalidomide.
8. Prior > or = to grade 3 (see Appendix III) allergic reaction/hypersensitivity to thalidomide.
9. Prior > or = grade 3 (see Appendix III) rash or any desquamating (blistering) rash while taking thalidomide.
10. Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation of study drug therapy.
11. History of cardiac disease, with New York Heart Association Class II or greater (see Appendix V).
12. Subjects who have received > 200mg/m2 of anthracycline or anthracendione either alone or in combination. (Additional caution must be taken in subjects with mediastinal radiation.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Study Completion 2007-06

PRIMARY OUTCOMES:
Phase I-To determine the maximum tolerated dose (MTD) and evaluate the safety profile of oral lenalidomide on days 1 - 21 and liposomal doxorubicin on day 1 every 28 days, as combination therapy to subjects with advanced ovarian or primary peritoneal ca
Phase II-To explore the anti-tumor activity of the combination of oral lenalidomide on days 1 - 21 and liposomal doxorubicin on day 1 every 28 days when given to subjects with advanced ovarian or primary peritoneal carcinoma.

SECONDARY OUTCOMES:
Phase I-To explore the anti-tumor activity of the combination of lenalidomide and liposomal doxorubicin when given to subjects with advanced ovarian or primary peritoneal carcinoma.
Phase II-To evaluate the safety profile of the combination of lenalidomide and liposomal doxorubicin when given to subjects with advanced ovarian or primary peritoneal carcinoma

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California at San Francisco, San Francisco, California
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - OU Health Sciences Center, Oklahoma City, Oklahoma
  - Swedish Cancer Institute, Seattle, Washington